CLINICAL TRIAL: NCT06875726
Title: Designing and Pilot Testing a Just-in-time Adaptive Intervention (JITAI) for Adolescent Depression Treatment in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Jenness, Assistant Professor: Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019936; R61MH132809 (NIH)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This is a single-arm study of a micro-randomized digital intervention for teens with depression. All teens will receive the intervention, and randomization of which time points a teen receives an intervention or not will occur within-subject. The intervention will consist of messages sent via a secure app. Intervention messages will be possible up to 2x/day with a 50% chance of being delivered at each time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Behavioral: Sidekick

INTERVENTIONS:
Behavioral: Sidekick — Sidekick is a just-in-time adaptive intervention that sends behavior change messages based on personalized sleep and physical activity goals.

SUMMARY:
The goal of this clinical trial is to learn if a tailored smartphone intervention called Sidekick can help improve sleep and physical activity for teenagers in depression treatment. The main question it aims to answer is:

Does Sidekick help teens improve sleep or physical activity?

Teen participants will be asked to complete surveys about how they are feeling and doing at the beginning of the study and throughout their participation. All teen participants will be able to use the Sidekick app during the study.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. 13 to 17 years old
3. PHQ-8 score ≥5
4. PHQ-8 rating of ≥1 on anhedonia, sleep, or fatigue items
5. Own a personal smartphone

Exclusion Criteria:

1. Active safety concerns (e.g., acute suicidal ideation)
2. Diagnosed developmental disability (e.g., autism spectrum)
3. Primary mental health diagnosis other than MDD according to baseline Mini-international Neuropsychiatric Interview (MINI) (comorbidity allowed when MDD primary)
4. Sleep disorder from another medical cause
5. Inability to engage in moderate exercise because of medical concerns;

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbance | Baseline to 4 weeks
  The PROMIS Sleep Disturbance 8a scale for adolescents is a self-report assessment of sleep difficulties over the past week. It includes 8 items related to sleep quality and disturbances rated on a 5-point scale. Raw scores (range: 8 - 40) are converted to normalized T-scores, with higher scores indicating greater sleep disturbance
Sleep related impairment | Baseline to 4 weeks
  The PROMIS Sleep-Related Impairment measure is a self-report assessment of the impact of sleep disturbances on daily functioning over the past week. It includes 8 items related to how sleep problems affect activities like school performance, mood, and social interactions, rated on a 5-point scale. Raw scores (range: 8-40) are converted to normalized T-scores, with higher scores indicating greater impairment in daily functioning due to sleep issues.
Sleep Quality | Baseline to 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report assessment of sleep quality over the past month. It includes 19 items covering sleep patterns, duration, disturbances, and daytime dysfunction. Response values are combined into components produce a global score (range: 0-21), with higher scores indicating poorer sleep quality and greater sleep-related difficulties.
Physical Activity Questionnaire - Adolescent | Baseline to 4 weeks
  The Physical Activity Questionnaire for Adolescents (PAQ-A) is a self-report assessment of physical activity levels in adolescents over the past 7 days. It includes 9 items related to the frequency and intensity of various physical activities, with responses on a 5-point scale. Scores are summed and averaged, with higher scores indicating greater physical activity levels.

SECONDARY OUTCOMES:
Depression | Baseline to 4 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report tool used to assess the severity of depressive symptoms over the past two weeks. It includes 9 items related to mood, interest, and other depressive symptoms, rated on a 4-point scale. Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms and greater impairment.
Anxiety | Baseline to 4 weeks
  The Generalized Anxiety Disorder-7 (GAD-7) is a self-report assessment of the severity of anxiety symptoms over the past two weeks. It includes 7 items related to anxiety-related feelings like worry, restlessness, and physical symptoms, rated on a 4-point scale. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms and greater impairment.

OTHER OUTCOMES:
Step Count | Baseline to 4 weeks
  Step count will be collected via the Garmin smartwatch. The average daily step count over the 2-week baseline data collection period will be compared to the average daily step count in the last week of the intervention.
Diagnostic Interview Schedule for Children | Baseline to 4 weeks
Activity Intensity | Baseline to 4 weeks
  Activity intensity will be collected via the Garmin smartwatch, categorized into light, medium, and vigorous. The average daily minutes of moderate + vigorous activity during the 2-week baseline data collection period will be compared to the average daily minutes of moderate + vigorous activity in the last week of the intervention.
Suicide Ideation | Baseline to 4 weeks
  The Suicide Ideation Questionnaire-Junior (SIQ-Jr) measures the frequency of suicide ideations in the past month. The 15-item self-report assessment records frequency on a 7 point scale ranging from "Almost every day" (0) to "I never had this thought" (7). Scores range from 0 to 90 with higher scores indicating greater frequency of SI.
Functional Impairment | Baseline to 4 weeks
  The Weiss Functional Impairment Rating Scale (WFIRS) is a self-report tool used to assess the functional impairment associated with ADHD symptoms across various domains, such as family, social, school/work, and emotional functioning. It includes 18 items rated on a 5-point scale. Total scores indicate the level of impairment, with higher scores reflecting greater functional difficulties and more significant impact on daily life.
Sleep Duration | Baseline to 4 weeks
  Sleep duration will be collected via the Garmin smartwatch. The average daily sleep duration (in minutes) during the 2-week baseline data collection period will be compared to the average daily sleep duration (in minutes) in the last week of the intervention.
Midpoint sleep variability | Baseline to 4 weeks
  The midpoint of sleep (clock time halfway between bedtime and waketime) will be collected via the Garmin smartwatch. The standard deviation of the midpoint during the two week baseline period will compared to the standard deviation of the midpoint during the last two weeks of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jenness, Ph.D., Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No